CLINICAL TRIAL: NCT04252313
Title: Music as an Adjunct to Combination Analgesia for Neonatal Circumcision: A Randomized Controlled Trial
Brief Title: Music as Analgesia During Neonatal Circumcision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Rana Sharara, Associate Professor of Clinical Pediatrics and Pediatric Critical Care, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: BIO-2018-0405
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Analgesia
Keywords: Music; Neonatal Circumcision
MeSH Terms: conditions — Agnosia | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either the control group [Only EMLA+Sucrose+Ring Block] or the Intervention [EMLA+Sucrose+Ring Block+ Music]
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The infant's parents signing the participation consent are blinded to the child's randomization allocation. The Surgeon performing the circumcision is wearing noise-cancelling headphones, therefore is unaware of the patient's randomization. The outcomes assessors are evaluating the videos in mute. Both surgeons and assessors are investigators on the study; only the statistician, the study coordinator and the assistant are aware of the randomization allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (No Intervention): This arm represents the control group. They will be undergoing the circumcision without any music, with the established standard for analgesia [EMLA+Sucrose+Ring Block]
- Group B: Music (Experimental): In addition to the standard analgesia as explained for group A, Music will be played from the "Baby Go to Sleep" playlist which includes nursery rhymes and lullabies metonymized to an actual human heartbeat (Houser, 1994). Music will start after the baby settles on the board and before the surgeon starts the procedure.
  Interventions: Other: Music

INTERVENTIONS:
Other: Music — Studies have been conducted to assess the effects of sound and noise on neonatal stress. Recently, music is being used in neonatal units to improve physiological and behavioral outcomes (Harling et al, 2009). Of the few studies done on the effectiveness of music during circumcision is a randomized double-blinded controlled trial conducted by Joyce et al (2001): it found that some physiologic outcomes were significantly lower among the music group in comparison to the EMLA group. They concluded that there is preliminary evidence to support the efficacy of EMLA and music in pain management of newborn circumcision; however, more rigorous studies are warranted for conclusive results.
  Arms: Group B: Music

SUMMARY:
Neonatal circumcision is one of the most frequently performed and more painful procedures. Sharara et al (2017) showed the combination of EMLA + Sucrose + Ring Block provides the highest standard of pain management. A combination which has been adopted by practitioners who perform circumcisions at the normal nursery at AUBMC. An element which is overlooked in its ability to enhance or suppress stress and consequently pain is sound/noise, music. The specific aim of this study is to test the added effectiveness of music (Group B: intervention) to the established standard for analgesia [EMLA + Sucrose + Ring Block] (Group A: control) in further managing the pain of newborn males undergoing circumcision.

DETAILED DESCRIPTION:
Scientific Context: Neonatal circumcision is one of the most frequently performed and more painful procedures. Sharara et al (2017) showed the combination of EMLA + Sucrose + Ring Block provides the highest standard of pain management. A combination which has been adopted by practitioners who perform circumcisions at the normal nursery at AUBMC. An element which is overlooked in its ability to enhance or suppress stress and consequently pain is sound/noise, music.

Hypothesis/Aims: The specific aim of this study is to test the added effectiveness of music (intervention) to EMLA + Sucrose + Ring Block (control group) in further managing the pain of newborn males undergoing circumcision.

Experimental design, subject selection/recruitment, procedures involving human subjects: A double blinded randomized controlled trial, comparing the control Group A to the intervention Group B: Music. All healthy, late pre-term and term (36-41 weeks) newborn males admitted to the normal nursery at the AUBMC whose parents request circumcision are eligible for recruitment following a negative auditory screening test. Following written consent from the parents, participants will be allocated to either control or intervention based on a prepared list of block randomization. Babies will be videotaped during the circumcision, legs and the field of operation will be excluded from view. This video will be evaluated by two blinded pediatricians using the validated Neonatal Infant Pain Scale/Score (NIPS).

4- Risks and Benefits, and Risk/Benefit Ratio: The risks are associated with the circumcision procedure itself, not the proposed intervention, these risks are rare and may include risks associated with the surgery, or adverse reactions to the pharmacological anesthetics administered. Benefits include maximal pain management. The ratio leans favorably towards the benefits.

Privacy and Confidentiality: All Co-investigators are blinded to the randomization. Babies will be marked as Baby 1, Baby 2, and Baby 3…etc. The videotaping will not include any identifying information, although the baby's face will be in view; the videos will be placed on a password protected IPad only used for the purposes of this study, in the study coordinator's possession, kept in a locked drawer. When evaluating these videos, the evaluators will view them on the IPad. No copies or duplicates will be made and shared, even among the team. The collected data will be coded and kept on a password protected computer, the coded file will be shared with the statistician for the purposes of analysis. Following IRB protocol, all study related materials will be destroyed and permanently deleted after 3 years from the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* All healthy, late pre-term and term (36-41 weeks) newborn males admitted to the normal nursery at the American University of Beirut Medical Center (AUBMC) who have successfully passed an auditory screening (including the AABR and/or OAE) and whose parents request circumcision are eligible for recruitment

Exclusion Criteria:

* Newborn males admitted to the normal nursery at the American University of Beirut Medical Center (AUBMC), who have not passed the auditory screening (including the AABR and/or OAE).

Ages: 24 Hours to 48 Hours | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — The study is about male neonatal circumcision.
Enrollment: 206 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale (NIPS) | 4-6 minutes. Change of the infants pain during Stage 1-6 of the circumcision.
  The NIPS is a non-intrusive, replicable, and objective tool for assessing pain responses. The tool uses five behavioral cues observed over time, with a composite score of 0 to 6, to determine the amount of pain or change in pain the infant is experiencing; scores more than 3 are indicative of pain.

SECONDARY OUTCOMES:
Heart Rate | 4-6 minutes. Change of the infants pain during Stage 1-6 of the circumcision.
  The infant is placed on a pulse oximeter during the circumcision to monitor his heart rate.
Oxygen Saturation | 4-6 minutes. Change of the infants pain during Stage 1-6 of the circumcision.
  The infant is placed on a pulse oximeter during the circumcision to monitor his oxygen saturation.
Crying Time | 4-6 minutes. Change of the infants pain during Stage 1-6 of the circumcision.
  The assistant will be timing the infant's crying during the circumcision, as an indicator of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Rana Sharara-Chami, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No
The data is only to be shared within the investigating team. The results will be shared in aggregate form.

REFERENCES:
- [Background] Lawrence J, Alcock D, McGrath P, Kay J, MacMurray SB, Dulberg C. The development of a tool to assess neonatal pain. Neonatal Netw. 1993 Sep;12(6):59-66. PMID 8413140
- [Result] Sharara-Chami et al. Combination Analgesia for Neonatal Circumcision: A Randomized Controlled Trial. Pediatrics. 2017;140(6):e20171935. Pediatrics. 2018 May;141(5):e20180500. doi: 10.1542/peds.2018-0500. Epub 2018 Apr 30. No abstract available. PMID 29712767
- [Derived] Sharara-Chami R, El-Hout Y, Lakissian Z, Hafez B, Abi-Gerges C, Fayad J, Charafeddine L, Tazian V, Tamim H, Zaghal A. Music as an adjunct to combination analgesia for neonatal circumcision: A randomized controlled trial. J Pediatr Urol. 2022 Apr;18(2):184.e1-184.e6. doi: 10.1016/j.jpurol.2021.12.011. Epub 2021 Dec 24. PMID 35000838